CLINICAL TRIAL: NCT00150631
Title: Danish Hypertension Prevention Project
Brief Title: Danish Hypertension Prevention Project - DHYPP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karin Skov (Other)
Collaborators: University of Aarhus (Other); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Karin Skov, consultant, ph.d., Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 20000114
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
Keywords: Hypertension; Prevention; Offspring; Prevent or delay development of hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active (candesartan) (Placebo Comparator): 12 mo treatment with candesartan
  Interventions: Drug: Candesartan
- placebo (Placebo Comparator): 12 mo placebo treatment

INTERVENTIONS:
Drug: Candesartan — placebo controlled double blind
  Other Names: atacand
  Arms: active (candesartan)

SUMMARY:
The present study examine healthy, normotensive subjects 18 to 36 years of age whose both parents have essential hypertension. The subjects receive treatment with either the AT1-antagonist candesartan cilexetil, 16 mg daily or placebo for one year. Then, treatment is withdrawn and the subjects is followed for 10 years to determine if the treatment has been able to either prevent or delay the development of hypertension. The primary objective is to determine whether pharmacological treatment with an angiotensin receptor blocker is able to restrain or delay the progression to hypertension. Secondary objectives are to investigate whether any long-term effect on blood pressure is related to the effect of treatment on renal haemodynamic function, or on the left ventricle mass.

DETAILED DESCRIPTION:
Essential hypertension, a major health problem worldwide, is a disease generally considered to require life-long treatment. However, evidence suggests that hypertension is caused by specific phenotypic changes caused by a combination of genetic and environmental factors. Thus, in principle, hypertension could be prevented by prevention of these phenotypic changes. Animal data indicate that early treatment that blocks the renin-angiotensin system have long-term effects after treatment withdrawal. The present human study is testing whether early treatment (with the AT1- antagonist) is able to have a persistent effect after stopping treatment.

This is a monocenter, double-blind, randomized, placebo-controlled study in healthy, normotensive (consultation diastolic blood pressure over 2 visits < 85 mmHg) subjects 18 to 36 years of age whose both parents have essential hypertension. The primary objective is to determine whether pharmacological treatment with an angiotensin receptor blocker is able to restrain or delay the progression to hypertension. Secondary objectives are to investigate whether any long-term effect on blood pressure is related to the effect of treatment on renal haemodynamic function, or on the left ventricle mass.

Subjects are recruited by use of hospital registers to identify persons who have received the indication essential hypertension, and are of an age that they may have children of the appropriate age. These persons are then mailed asking if they do have children with a partner who is also hypertensive, and asking permission to contact the children. The diagnosis of hypertension of the parents is checked following evaluation by the physicians who are treating them.

One hundred subjects were randomly assigned to one of two treatment groups: placebo; or candesartan cilexetil, 16 mg, once daily. Before inclusion and after 12 months of treatment glomerular filtration rate, renal vascular resistance, echocardiography and 24-hour blood pressure monitoring were performed. Subjects were evaluated at 0.5, 1, 2, 4, 6 and 10 months to ensure compliance and to control blood pressure. After 12-months of treatment, 24-hour blood pressure monitoring were performed in a scheduled manner over a 10-year period. The primary effect parameter is 24-hour blood pressure measured 10 years after withdrawal of treatment. Interim analyses will be made at 1, 2 and 5 years by an independent data committee. Secondary effect parameters will be numbers on antihypertensive treatment at 2, 5 and 10 years after withdrawal, as well as the effect of treatment on renal vascular resistance and left ventricular mass.

A substudy is comparing renal haemodynamics and genetic profil of the subjects with persons having normotensive parents.

ELIGIBILITY:
Inclusion Criteria:

1. Both parents have essential hypertension
2. Age 18 - 36 years
3. Caucasians
4. Diastolic blood pressure less than 85 mmHg at inclusion time
5. Female participants using orale anticonceptives ot intrauterine devices

Exclusion Criteria:

1. Clinical or biochemically signs of disease in kidney, liver, or endocrine organs
2. Diastolic blood pressure above 85 mmHg at inclusion time
3. Pregnancy or pregnancy wish
4. Daily medication, except for orale anticoncetives -

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2000-11; Primary Completion 2004-01 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to determine whether pharmacological treatment with an angiotensin receptor blocker is able to restrain or delay the progression to hypertension. | 10 years
Secondary outcomes are to investigate whether any long-term effect on blood pressure is related to the effect of treatment on renal haemodynamic function, or on the left ventricle mass. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: michael mulvany, prof, Study Chair — Dept. of Pharmacology, Aarhus University
Locations (1):
- Karin Skov, Aarhus, Denmark